CLINICAL TRIAL: NCT00589719
Title: Asthma in the Delta Region of Arkansas (ADRA): Prevalence and Morbidity
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Dr. Tamara Perry, University of Arkansas for Medical Sciences
Other Study IDs: 39931
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Asthma
Keywords: Asthma; minority; low-income; African American; Arkansas
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2000,3000,4000: Children at risk for asthma were identified using a cross-sectional asthma screening survey.

SUMMARY:
The purpose of the study is to conduct a cross-sectional study to examine asthma prevalence and morbidity in a predominately minority, low-income population in rural Arkansas.

DETAILED DESCRIPTION:
Asthma is the leading chronic disease of childhood in the United States and an important public health concern in Arkansas. Arkansas, a predominately rural state, has one of the leading mortality rates in the nation for African Americans. The specific aims of the study will examine asthma prevalence in children age 4-17 years old in public schools in Eudora and Marvell Arkansas. The study will also examine asthma morbidity among identified asthmatics by characterizing activity limitation, days missed from school, daytime and nocturnal symptoms, healthcare utilization and medication use. The specific aims of the current study will provide novel data on an understudied population of asthmatics and will test our working hypotheses that pediatric asthma prevalence in the Delta region of Arkansas is higher than national estimates; and asthma diagnosis is related to significant morbidity among rural asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-17 years, enrolled in the public schools in Eudora and Marvell Arkansas.

Exclusion Criteria:

* Children aged 18 or older enrolled in the public schools in Eudora and Marvell Arkansas were excluded.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: During the 2005-2006 school year, primary caregivers of all students aged 4-17 years attending public school in Eudora and Marvell Arkansas were asked to complete an asthma screening survey regarding their child. The schools are located in two non-contiguous counties in the Delta region of Arkansas and are in rural low-income areas of the state where more than one-third of families with children 5-17 years old meet the 2000 poverty line (Census bureau).
Sampling Method: Non-Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2005-08; Primary Completion 2006-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The findings suggest that asthma diagnosis and active symptoms are prevalent among this predominately minority and low-income rural population in the Arkansas region of the Mississippi Delta. | One year

SECONDARY OUTCOMES:
High rates of inadequately controlled asthma are evidenced by activity limitation, medication use and increased healthcare utilization. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Galant SP, Crawford LJ, Morphew T, Jones CA, Bassin S. Predictive value of a cross-cultural asthma case-detection tool in an elementary school population. Pediatrics. 2004 Sep;114(3):e307-16. doi: 10.1542/peds.2003-0575-F. PMID 15342891